CLINICAL TRIAL: NCT03377777
Title: Development of Infants and Young Children Living in the Amazon Region of Peru: Relationship With Anemia, Chronic Malnutrition, and Gut Microbiota.
Brief Title: The Effect of Anemia in Infancy on the Microbiome and Systemic Metabolism
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: Universidad Peruana Cayetano Heredia (Other); Asociacion Civil Selva Amazonica (Other)
Responsible Party: Sponsor
Other Study IDs: GAIN08112014; 00000000 (Other: UCDavis IRB exempt)
Record Dates: First submitted 2017-12-11; First posted 2017-12-19 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Anemia; Iron-deficiency; Iron Deficiency Anemia
Keywords: Anemia; Iron-deficiency; Iron-deficiency anemia; Infants; Metabolomics; Microbiome
MeSH Terms: conditions — Anemia; Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infants: Outwardly healthy male and female infants at 6-7 months or 12-13 months. No intervention.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
Serum and fecal samples were collected from infants at either 6-7 m of age or 12-13 m of age. Serum and feces were analyzed locally for hemoglobin status or evidence of parasites, and standard of care was provided. Excess serum was transported to UC Davis for metabolomics analysis and the University of Hohenheim for iron status assessment and measurement of inflammatory markers. Fecal samples were transported to UC Davis for measurement of the microbiome structure and function.

DETAILED DESCRIPTION:
Sample collection occurred between August and November 2014. A total of 203 infants and their parents (101 at 6-7 m of age and 102 at 12-13 m of age) receiving care at the Moronacocha Health Center in Iquitos, Peru were recruited. All subjects were residents of Moronochocha, Iquitos, Loreto, outwardly healthy, and born at term with a birth weight of at least 2,500 g. Venous blood samples were collected by a lab technician at the local health center. Hemoglobin concentrations were immediately measured, and treatment given if warranted. Samples were subsequently transported to Selva Amazonica clinic, centrifuged, and serum was stored at -80 °C. Stool samples were collected by caregivers from diapers at home, taken to Selva Amazonica Clinic, and aliquoted. Fecal samples were analyzed for parasites at Selva Amazonica, and any necessary treatment was provided at the local health center. Serum and stool samples were shipped to UC Davis on dry ice, where they were stored at -80 °C until metabolomics and microbiome analyses. Serum aliquots were also shipped to the University of Hohenheim, Stuttgart, Germany for iron assessment, and measurement of inflammatory markers. All data integration and interpretation was performed at UC Davis.

ELIGIBILITY:
Inclusion Criteria:

* Outwardly healthy,
* birthweight > 2,500 g
* term births
* residents in Moronacocha, Iquitos, Loreto

Exclusion Criteria:

* Obvious signs of illness or malnutrition
* birthweight < 2,500 g
* preterm birth
* not a resident of Moronacocha, Iquitos, Loreto

Ages: 6 Months to 13 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Outwardly healthy 6-7 month, and 12-13 month male and female infants born at term with a birthweight > 2,500 g.
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2014-11-30 (Actual); Study Completion 2014-11-30 (Actual)

PRIMARY OUTCOMES:
Anemia status | 6-7 months or 12-13 months
  Anemia status [Hb] ≤ 110 g/L

IPD SHARING:
Plan to Share IPD: Yes
Microbiome sequencing data will be shared in a public repository (with iron status included as meta data).
Time Frame: Once study has been published
Access Criteria: Publicly available

REFERENCES:
- [Derived] McClorry S, Zavaleta N, Llanos A, Casapia M, Lonnerdal B, Slupsky CM. Anemia in infancy is associated with alterations in systemic metabolism and microbial structure and function in a sex-specific manner: an observational study. Am J Clin Nutr. 2018 Dec 1;108(6):1238-1248. doi: 10.1093/ajcn/nqy249. PMID 30351381